CLINICAL TRIAL: NCT05021575
Title: Effects of COVID-19 Pandemic on Personal and Public Health and Functioning of Health Care System: Case Study of the CirculatORy System in LiThuania
Brief Title: Effects of COVID-19 Pandemic on a Health Care System: Case Study of the CirculatORy System in LiThuania
Acronym: COVID-COR-LT
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: Institute of Hygiene, Lithuania (Unknown); National Health Insurance Fund under the Ministry of Health, Lithuania (Unknown); Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Jelena Čelutkienė, Senior Researcher and Professor in Clinic of Cardiac and Vascular Diseases, Centre of Cardiology and Angiology, Vilnius University; Senior cardiologist in Unit of Stress testing, Vilnius University Hospital Santaros Klinikos, Vilnius University
Other Study IDs: S-COV-20-27; S-COV-20-27 (Other Grant/Funding Number: Research Council of Lithuania); 2020/8-1247-730 (Other: Lithuanian Bioethics Commitee)
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular diseases; COVID-19; health care system; cardiovascular mortality; hospitalizations; outpatient care; cardiovascular interventions
MeSH Terms: conditions — Cardiovascular Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2020: Data on outpatient care, hospitalisation and cardiovascular mortality were collected for the year 2020.
  Interventions: Other: Data collection on outpatient care; Other: Data collection on hospitalisation; Other: Data collection on cardiovascular mortality; Other: Data collection of patients presenting to the tertiary care centre with acute coronary syndrome
- 2019: Data on outpatient care, hospitalisation and cardiovascular mortality were collected for the year 2019.
  Interventions: Other: Data collection on outpatient care; Other: Data collection on hospitalisation; Other: Data collection on cardiovascular mortality; Other: Data collection of patients presenting to the tertiary care centre with acute coronary syndrome

INTERVENTIONS:
Other: Data collection on outpatient care — Outpatient data from 1 January to 30 November of the analysed year were obtained from National Health Insurance Fund under the Ministry of Health.
  Outpatient data related to cardiovascular diseases (CVD) were collected as described:
  1. data on visits were collected using ICD-10 codes I00-I99 and other CVD related codes (e.g., certain Z, Q codes, J81.0, R57.0)
  2. data were collected from CVD prevention program
  3. data on interventional cardiology were collected from day care facility regardless of the diagnosis.
  Date of the visit, patient age, sex and municipality, service level (primary, secondary or tertiary), type of service and main diagnosis were recorded.
Other: Data collection on hospitalisation — Hospitalisation data from 1 January to 30 November of the analysed year were obtained from National Health Insurance Fund under the Ministry of Health.
  Data on hospitalisation were collected if any of the diagnoses (principal or secondary) were in I00-I99 range. Hospitalisation data covered hospitalisation date, patient age, sex, municipality and outcome. Data on cardiovascular procedures performed during hospitalisations included date of the procedure and ACHI (Australian Classification of Health Interventions) code.
Other: Data collection on cardiovascular mortality — Data on cardiovascular mortality were obtained from death certificates provided by Causes of Death Registry from Institute of Hygiene and covered the period from 1 January to 31 December of the analysed year. Death certificates were included in the study when cause of death was adjudicated to be in I00-I99 range. Date and place of death (hospital, home, other or unspecified), patient age and sex were recorded.
Other: Data collection of patients presenting to the tertiary care centre with acute coronary syndrome — Demographic, clinical and percutaneous coronary intervention (PCI) related data were collected from 1st March to 30th June of the analysed year. The timing of the chest pain onset, call for medical help, first medical contact (FMC), arrival to PCI centre, and PCI procedure were analysed.

SUMMARY:
Coronavirus disease of 2019 (COVID-19) affected the health care systems all around the world. The collateral damage of the pandemic on the cardiovascular (CV) care and CV mortality has been noticed and reported early. In Lithuania, first quarantine measurements were introduced on 16th March and lifted on 16th June of 2020, limiting contact appointments to urgent care only. This led to a substantial proportion of routine cardiovascular appointments, diagnostic and therapeutic procedures being cancelled and greatly limited the availability of cardiovascular care. The prognostic impact of this has not been appropriately analysed. Also, comprehensive analyses of the changes in national CV services, including outpatient care and hospitalisations and CV mortality, during different periods of the pandemic (during first and second waves and in between) are scarce. The objectives of this population-based study were: (1) to assess the impact of the COVID-19 pandemic on CV care (2) to compare rates of outpatient care visits and hospitalisations of cardiovascular patients in different periods of 2019 and 2020 (3) to compare the rates of CV mortality in Lithuania in different periods of 2019 and 2020 (4) to investigate sex and age differences in CV care and CV mortality

DETAILED DESCRIPTION:
COVID-19 pandemic has greatly affected the world and changed health care in almost every country. During the spring of 2020, first pandemic wave was of different scale in different countries. In countries affected by the virus the most, a majority of the studies focused on the direct impact of COVID-19 on community health. It was noticed promptly that the novel virus is especially high-risk for patients with cardiovascular comorbidities. Furthermore, the collateral damage of COVID-19 pandemic on the provision of cardiovascular (CV) care and cardiovascular mortality was also reported early in several nationwide and selected cohort studies. The research was mostly focused on acute cardiovascular conditions; changes in hospital admissions and early mortality after myocardial infarction were also often analysed. Meanwhile, a substantial proportion of routine appointments, diagnostic and therapeutic procedures was cancelled. Data on the changes in total national CV services, including out- and in-patient health care facilities, acute and chronic conditions, during the outbreak, between the two pandemic waves and onwards are scarce. First case of COVID-19 in Lithuania was confirmed on 28th February 2020. First nationwide quarantine was introduced by Lithuanian government on 16th March and ended on 16th June. In that period, although Lithuania was reported among the least affected countries according to World Health Organization - 1 773 COVID-19 cases were recorded and 86 patients (of whom 10 patients died from other causes after testing positive for SARS-CoV-2) had died before the end of quarantine, Lithuanian government limited contact appointments to urgent conditions only. The utmost efforts to provide triage, follow-up care by telephone call and e-prescriptions were recommended. This greatly affected availability of cardiovascular care. The second pandemic wave in Lithuania was substantially more severe. Consequently, the second nationwide quarantine was implemented on 7th November, 2020. Contact appointments were not limited by the government; however, the scope of CV care was again negatively affected, mostly by the strained health care system.

We analysed the indirect impact of the COVID-19 pandemic in a country, which was hit by two very different pandemic waves. The objectives of this population-based study were: (1) to assess the impact of the COVID-19 pandemic on CV care (2) to compare rates of outpatient care visits and hospitalisations of cardiovascular patients in different periods of 2019 and 2020 (3) to compare the rates of CV mortality in Lithuania in different periods of 2019 and 2020 (4) to investigate sex and age differences in CV care and CV mortality

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old adult patients
* Included in either National Health Insurance Fund outpatient and hospitalisation registries related to cardiovascular diseases from 1st January 2019 to 30th November 2020
* Included in Causes of Death Registry from Institute of Hygiene with cardiovascular diagnoses from 1st January 2019 to 31st December 2020.

Exclusion Criteria:

* Cases, when sex was not available were excluded from sex differences analysis.
* Death certificates where place of death was unspecified were excluded from death place analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) included in either National Health Insurance Fund outpatient and hospitalisation registries related to cardiovascular diseases from 1st January 2019 to 30th November 2020 or in Causes of Death Registry from Institute of Hygiene with cardiovascular diagnoses from 1st January 2019 to 31st December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 839678 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of outpatient care visits for cardiovascular reasons in Lithuania in 2019 and 2020 | 2 years
  Assessing the impact of the COVID-19 pandemic on provision of CV care at the national and regional level in Lithuania
Number of cardiovascular hospitalisations in Lithuania in 2019 and 2020 | 2 years
  Assessing the impact of the COVID-19 pandemic on provision of CV care at the national and regional level in Lithuania
Cardiovascular mortality rates in Lithuania in 2019 and 2020 | 2 years
  Assessing the impact of the COVID-19 pandemic on provision of CV care at the national and regional level in Lithuania

SECONDARY OUTCOMES:
Evaluation of sex and age differences in changes of CV care provision and CV deaths during the pandemic and comparison between 2019 and 2020 | 2 years
  Comparison of cardiovascular outpatient care visits, hospitalisation numbers and cardiovascular mortality rates between men and women and between different age groups.
In-hospital mortality rates in Lithuania in 2019 and 2020 | 2 years
  Comparison of mortality rate in hospitalised patients in Lithuania between 2019 and 2020
Comparison of distribution of death places in Lithuania in 2019 and 2020 | 2 years
  Assessing the differences in the death places written in the death certificates of the people deceased from cardiovascular causes between 2019 and 2020
Comparison of all-cause mortality during the hospital stay and at 3 months of follow-up in patients presenting to a tertiary care centre with acute coronary syndrome during the first quarantine in 2020 and in a corresponding period of 2019 | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- Lithuania (3):
  - Institute of Hygiene, Vilnius
  - National Health Insurance Fund under the Ministry of Health, Lithuania, Vilnius
  - Vilnius University, Vilnius

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celutkiene J, Cerlinskaite-Bajore K, Bajoras V, Visinskiene R, Lizaitis M, Budrys P, Buivydas R, Gurevicius R, Serpytis P, Davidavicius G. Collateral effect of the COVID-19 pandemic on cardiology service provision and cardiovascular mortality in a population-based study: COVID-COR-LT. Clin Res Cardiol. 2022 Oct;111(10):1130-1146. doi: 10.1007/s00392-022-02033-y. Epub 2022 May 12. PMID 35552504